CLINICAL TRIAL: NCT00989183
Title: Lifestyle Factors and Their Impact on Ovarian Reserve
Brief Title: Lifestyle Factors Study
Status: Completed | Type: Observational
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 1964
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Reproductive Age; Oophorectomy for Benign Indications
Keywords: Ovaries; Reproductive Age; Oophorectomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Telomere length assay
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Women undergoing a bilateral or unilateral oophorectomy at OU Medical Center, Oklahoma City, Oklahoma — Women undergoing an elective bilateral or unilateral oophorectomy at OU Medical Center, Oklahoma City, Oklahoma Age range 21-55 years old

SUMMARY:
The goals of this research proposal are to further our understanding of the reproductive aging process in women and to improve our ability to clinically assess and model reproductive aging. Reproductive aging is a continuous process that begins many years prior to menopause. Women in their late 30s and early 40s usually maintain normal menstrual function and ovulatory status, yet fertility in these women is considerably compromised compared to younger women. The primary mechanism of reproductive aging is through the process of ovarian primordial follicle (egg) depletion, a process that exhibits considerable variation between women. As a result, the age at which an individual begins to experience infertility and menstrual cycle changes secondary to follicle depletion also varies significantly and is difficult to predict. Multiple studies have investigated the impact of lifestyle choices (tobacco use, oral contraceptives, BMI, alcohol use, and parity) on reproductive lifespan by correlating the impact of these exposures with the age of spontaneous menopause. Although occasionally in agreement, many of these studies report contradictory findings. Alcohol use either delays or has no effect upon the age of spontaneous menopause. Similarly, oral contraceptive pill use has been suggested to both accelerate and delay the onset of menopause. The most consistent findings regarding the impact of these factors is an acceleration in the age of menopause by 1-2 years in smokers. Given the lack of consistent findings in these investigations, the exact impact of lifestyle factors on reproductive age is currently unknown. Nevertheless, the magnitude of such exposures in the U.S. population is considerable, with 19% of adult women using oral contraceptives and 19.2% current smokers according to recent statistics. This proposal seeks to develop better models of normal female reproductive aging through anatomical studies investigating the impact of lifestyle choices on ovarian primordial follicle number. A secondary aim is to determine the relationship between newly described markers developed to assess biological aging in other organ systems (white blood cell telomere length and the measurement of advanced glycation end products (AGEs) through skin autofluorescence) and reproductive age.

DETAILED DESCRIPTION:
In order to test the hypotheses, we will obtain whole ovaries (single or pairs) from 65 healthy females between the ages of 21 and 55 undergoing surgical oophorectomy at OU Medical Center for benign indications.

* informed consent
* collection of baseline demographic data (height, weight, ethnicity, age)
* completion of structured interview to obtain information regarding oral contraceptive, ethanol, tobacco use and socioeconomic status
* Measurements of FSH, estradiol, inhibin B, AMH, white-blood cells for telomere length, measurement of hemoglobin A1C to control for blood glucose levels
* AFC as determined by transvaginal ultrasound exam
* skin autofluorescence measurement
* subjects then undergo surgery with their primary care gynecologist
* determination of ovarian PF number by modern morphometric methods

ELIGIBILITY:
Inclusion Criteria:

* Undergoing gynecologic operations in which a bilateral or unilateral oophorectomy is performed at OU Medical Center, Oklahoma City
* 21-55 years old

  * NOTE: Must be willing to travel to Oklahoma City to participate. Need to have the transvaginal ultrasound and skin autofluorescence measurement at the OU Physicians Reproductive Health Clinic in Oklahoma City, Oklahoma.

Exclusion Criteria:

* Gynecological malignancy
* Chemotherapy or radiation treatment
* Autoimmune disease
* Prior ovarian surgery
* Subjects with ovarian pathology such as polycystic ovaries, endometrioma, dermoid

Ages: 21 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: We will obtain whole ovaries (single or pairs) from 65 healthy females between the ages of 21 and 55 undergoing surgical oophorectomy for benign indications at the OU Medical Center, Oklahoma City, Oklahoma.
  *NOTE: Must be willing to travel to Oklahoma City to participate. Need to have the transvaginal ultrasound and skin autofluorescence measurement at the OU Physicians Reproductive Health Clinic in Oklahoma City, Oklahoma.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2009-08-19 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
To determine the impact of lifestyle choices (body-mass index, smoking, oral contraceptive use, and ethanol use) on ovarian primordial follicle (PF) number with the goal of incorporating these parameters into our model of reproductive aging in women. | 2 years

SECONDARY OUTCOMES:
Determine whether white blood cell telomere length and AGE measured by skin autofluorescence are correlated with ovarian PF number. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Karl R Hansen, MD, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States